CLINICAL TRIAL: NCT02275208
Title: A Prospective, Multi-center, Single-arm Study of the Stomach, Intestinal and Pylorus Sparing (SIPS) Procedure
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVSIPS0447
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: SIPS the stomach, intestinal, pylorus, sparing procedure — Bariatric Procedure

SUMMARY:
This study is a prospective, multi-center, single-arm study evaluating the SIPS procedure. Subjects who meet the eligibility criteria will be considered for study participation and will be followed through 12 months.

DETAILED DESCRIPTION:
SIPS is a single-anastomosis duodeno-intestinal switch procedure. Preliminary data from Sanchez-Pernaute et al. (Surg Obes Relat Dis 2013;9:731) indicates that this procedure is safe, quick to perform, and offers good results for treatment of both morbid obesity and its metabolic comorbidities. CovidienTM plans to further investigate this procedure and has proposed a prospective clinical study to obtain data on subject outcomes through 12 months following the SIPS procedure.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18-65 years of age
* The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent
* The subject is under consideration for surgery for obesity or metabolic disease and elects to undergo a primary SIPS procedure
* The subject has a BMI of 35-40 kg/m2 with at least 1 obesity-related comorbidity or a BMI of 40-60 kg/m2

Exclusion Criteria:

* Any female subject who is pregnant, or is actively breast-feeding
* Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those with psychological concerns or those without sufficient mental capacity)
* The procedure is an emergency procedure
* The procedure is a revision/reoperation for the same indication
* The subject is unable or unwilling to comply with the study requirements or follow-up schedule
* The subject has conditions which, in the opinion of the investigator, will not be appropriate for the study (e.g. severe cardiovascular disease, history of gastrointestinal (GI) malignancy, history of upper GI surgery, open cholecystectomy, history of intestinal surgery, immunosuppression, or non-ambulatory)
* The subject has an estimated life expectancy of less than 6 months
* The subject has participated in an investigational drug or device research study within 30 days of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multi-center, single-arm study. Patients who have elected to undergo bariatric surgery using the SIPS procedure (according to patient and investigator assessment and standard of care) will be evaluated for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is excess weight loss (EWL) at 12 months. | 12 months

SECONDARY OUTCOMES:
SIPS-related adverse events at all timepoints | 12 months
Resolution of comorbidities at 1, 6, and 12 months | 12 months
Quality of life (QOL) (SF-36 and gastroesophageal reflux disease - health related quality of life [GERD-HRQL]) at 6 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Parker, Colorado
  - Florida Hospital Celebration Health, Celebration, Florida
  - Mount Kisco, New York
  - New York, New York
  - Cary, North Carolina
  - Durham, North Carolina
  - Salt Lake City, Utah